CLINICAL TRIAL: NCT01162655
Title: Delivery of Cognitive-Behavioral Treatment for Insomnia Via Telehealth or Internet
Brief Title: Cognitive-Behavioural Therapy (CBT) for Insomnia Via Internet or Telehealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Health Sciences Centre Foundation, Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Maxime Holmqvist, Clinical Psychologist & Assistant Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H2009:110
Record Dates: First submitted 2009-12-22; First posted 2010-07-14 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Insomnia
Keywords: Insomnia; Cognitive-Behavioral Therapy; Internet; Telehealth
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telehealth (Experimental): Complete CBT group via telehealth
  Interventions: Behavioral: Cognitive-behavioral therapy for Insomnia (CBT)
- Internet (Experimental): Complete Internet-based CBT program
  Interventions: Behavioral: Cognitive-behavioral therapy for Insomnia (CBT)

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy for Insomnia (CBT) — 6-week course of CBT delivered either using internet or telehealth

SUMMARY:
Cognitive-Behavioural Therapy (CBT) is an effective treatment for chronic insomnia, which is a prevalent and costly problem. This pilot study will compare the effectiveness of two brief (6 week) psychological interventions delivered to residents of rural Manitoba using Telehealth or an interactive Internet-based platform. It is hypothesized that a) participants in the Telehealth condition will report significantly greater improvements in sleep parameters(e.g., sleep efficiency, time awake in bed, sleep-onset latency),insomnia severity, and daytime fatigue than those in the Internet condition and that b)participants in the Telehealth condition will show better adherence to treatment and greater satisfaction with treatment than those in the Internet condition.

ELIGIBILITY:
Inclusion Criteria:

* Must be residents of rural Manitoba (Canada)
* Must meet research diagnostic criteria for insomnia
* Must have access to a computer and high-speed internet

Exclusion Criteria:

* Comorbid conditions (medical and psychiatric) must be stable

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2010-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity | 6 weeks
  The primary outcome measure will be insomnia severity, as assessed by the Insomnia Severity Index (ISI; Morin, 2003), a 6-item self-report measure of impairment due to sleep difficulties

SECONDARY OUTCOMES:
Sleep diary data | 6 weeks
  Sleep diaries are a standard daily outcome measure for insomnia. The version used here (Morin, 1993) includes information regarding total sleep time, sleep-onset latency, sleep-efficiency, number of night awakenings, time awake in then night, sleep quality, and frequency of use of sleep medications.

CONTACTS AND LOCATIONS:
Overall Officials: Maxine Holmqvist, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Centre, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Holmqvist M, Vincent N, Walsh K. Web- vs. telehealth-based delivery of cognitive behavioral therapy for insomnia: a randomized controlled trial. Sleep Med. 2014 Feb;15(2):187-95. doi: 10.1016/j.sleep.2013.10.013. Epub 2013 Dec 31. PMID 24461370